CLINICAL TRIAL: NCT05049226
Title: A Randomized, Observer-blind Trial to Assess the Immunogenicity and Safety of Third Dose Vaccination With AstraZeneca COVID-19 Vaccine or Pfizer/BioNTech COVID-19 Vaccine Among Thai Adults Receiving Two Doses of Sinovac
Brief Title: Third Dose Vaccination With AstraZeneca or Pfizer COVID-19 Vaccine Among Adults Received Sinovac COVID-19 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Clinixir Co., Ltd. (Unknown); Program Management Unit-C (PMU-C), governed by Ministry of Higher Education, Science, Research and Innovation (MHESI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TVTN001
Record Dates: First submitted 2021-09-14; First posted 2021-09-20 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Infection; COVID-19 VACCINE
Keywords: COVID-19 Infection; COVID-19 Respiratory Infection; COVID-19 VACCINE; AstraZeneca COVID-19 VACCINE; AstraZeneca COVID-19 (ChAdOx1 AZD1222) vaccine; Pfizer/BioNTech COVID-19 VACCINE; Pfizer/BioNTech COVID-19 (BNT162b2) vaccine; Thai adults; full dose AstraZeneca COVID-19 VACCINE; half dose AstraZeneca COVID-19 VACCINE; full dose Pfizer/BioNTech COVID-19 VACCINE; half dose Pfizer/BioNTech COVID-19 VACCINE; Sinovac COVID-19 Vaccine; immunogenicity; safety
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Unblinded study staff will be responsible for preparing study products (in accordance with the randomly determined assignment), administering the study vaccine, and handling all drug accountability procedures. These personnel will not participate in the other aspects of the clinical trial, to help ensure the integrity of the blind at the site. Unblinded staff will retrieve a participant's randomization assignment after being informed by the PI or designee that a participant is eligible for randomization. They will prepare study vaccine (AZ or PF) with dose (full or half dose) based on the participant's randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two doses of SV at interval 60 to less than 90 days (Experimental): Participants who have received two doses of SV at interval 60 to less than 90 days
  Interventions: Biological: AstraZeneca ChAdOx1 AZD1222 vaccine (AZ) full dose; Biological: Pfizer/BioNTech BNT162b2 vaccine (PF) full dose; Biological: AstraZeneca ChAdOx1 AZD1222 vaccine (AZ) half dose; Biological: Pfizer/BioNTech BNT162b2 vaccine (PF) half dose
- Two doses of SV at interval 90 to less than 120 days (Experimental): Participants who have received two doses of SV at interval 90 to less than 120 days
  Interventions: Biological: AstraZeneca ChAdOx1 AZD1222 vaccine (AZ) full dose; Biological: Pfizer/BioNTech BNT162b2 vaccine (PF) full dose; Biological: AstraZeneca ChAdOx1 AZD1222 vaccine (AZ) half dose; Biological: Pfizer/BioNTech BNT162b2 vaccine (PF) half dose
- Two doses of SV at interval 120 to 180 days (Experimental): Participants who have received two doses of SV at interval 120 to 180 days
  Interventions: Biological: AstraZeneca ChAdOx1 AZD1222 vaccine (AZ) full dose; Biological: Pfizer/BioNTech BNT162b2 vaccine (PF) full dose; Biological: AstraZeneca ChAdOx1 AZD1222 vaccine (AZ) half dose; Biological: Pfizer/BioNTech BNT162b2 vaccine (PF) half dose

INTERVENTIONS:
Biological: AstraZeneca ChAdOx1 AZD1222 vaccine (AZ) full dose — Astrazeneca COVID-19 (ChAdOx1 AZD1222) vaccine:
  One dose (0.5 ml) contains: COVID-19 Vaccine (ChAdOx1-S* recombinant) 5 × 10^10 viral particles (vp)
  *Recombinant, replication-deficient chimpanzee adenovirus vector encoding the SARS-CoV-2 Spike glycoprotein. Produced in genetically modified human embryonic kidney (HEK) 293 cells.
  Administer: Intramuscular (IM) injection in the deltoid muscle
Biological: Pfizer/BioNTech BNT162b2 vaccine (PF) full dose — Pfizer-BioNTech COVID-19 (BNT162b2) vaccine:
  Diluent: 0.9% sodium chloride (normal saline, preservative-free)
  Administer: Intramuscular (IM) injection in the deltoid muscle
Biological: AstraZeneca ChAdOx1 AZD1222 vaccine (AZ) half dose — Astrazeneca COVID-19 (ChAdOx1 AZD1222) vaccine:
  One dose (0.5 ml) contains: COVID-19 Vaccine (ChAdOx1-S* recombinant) 5 × 10^10 viral particles (vp)
  *Recombinant, replication-deficient chimpanzee adenovirus vector encoding the SARS-CoV-2 Spike glycoprotein. Produced in genetically modified human embryonic kidney (HEK) 293 cells.
  Administer: Intramuscular (IM) injection in the deltoid muscle
Biological: Pfizer/BioNTech BNT162b2 vaccine (PF) half dose — Pfizer-BioNTech COVID-19 (BNT162b2) vaccine:
  Diluent: 0.9% sodium chloride (normal saline, preservative-free)
  Administer: Intramuscular (IM) injection in the deltoid muscle

SUMMARY:
This prospective, multi-center, randomized, observer-blind Phase 2 study. A total of 1320 participants will be divided into 2 groups (660 each) receiving either full dose or half dose of either AZ or PF.

Each group is further stratified into 3 subgroups according to three interval duration in term of days after second dose of SV for 60 to less than 90 days, 90 to less than120 days and 120 to 180 days. Each group will be randomized to receive either AZ or PF in 1:1 ratio.

Subjects who fulfilled eligibility criteria will be randomly assigned to receive either full dose or half dose of AZ or PF in 1:1 ratio as an IM injection in the deltoid muscle at Visit 1 (V1). Subjects will be follow-up for assessing immunity at day 28 (V3), day 60 (V4) and day 90 (V5) and for safety at day 7 (V2), day 28 (V3), day 60 (V4) and day 90 (V5). At least 50% from each subgroup will be randomly selected to provide additional blood at baseline (V1, day 0) and day 28 (V3) to be used for assessment of T-cell-mediated immunity (CMI)

DETAILED DESCRIPTION:
This study has been designed to assess immune response and safety of third dose vaccination with AstraZeneca ChAdOx1AZD1222 vaccine or Pfizer/BioNTech BNT162b2 vaccine among Thai subjects who have received two doses of Sinovac.

The types of vaccines provided by the government included 7.7 million doses of inactivated vaccine manufactured by Sinovac and 6.5 million doses of AstraZeneca ChAdOx1 AZD1222 vaccine.

With the limited supplies of COVID vaccines in many regions of the world especially in LMIC including Thailand and the evidences of waning immunity of especially inactivated vaccine have raised the concerns whether third dose is needed.

The third dose that available now in Thailand are AstraZeneca ChAdOx1AZD1222 vaccine (AZ)/ Pfizer/BioNTech BNT162b2 vaccine (PF) and whether this can be provided with half dose so that the vaccination coverage is going to be higher in spite of limited vaccine supplies.

A number of studies have proved that COVID-19 vaccines are effective at preventing people from getting severe COVID-19 disease. However, the vaccines do not only reduce the chance of infection, but they also help to mitigate disease severity.

Study population: Male and female adults aged equal or more than 20 years who received two doses of Inactivated COVID-19 vaccine developed by Sinovac (given at 21-28 days apart) at different intervals of 60 to less than 90 days, 90 to less than120 days and 120 to 180 days

This prospective, multi-center, randomized, observer-blind Phase 2 study, A total of 1320 participants will be divided into 2 groups (660 each) receiving either full dose or half dose of either AZ or PF.

Each group is further stratified into 3 subgroups according to three interval duration in term of days after second dose of SV for 60-less than 90 days, 90-less than120 days and 120-180 days respectively. Subjects who fulfilled eligibility criteria will be randomly assigned to receive either full dose or half dose of AZ or PF in 1:1 ratio as an IM injection in the deltoid muscle at Visit 1 (V1).

All participants will be randomized based on dose given either full dose or half dose and further stratify accordingly by Interactive web-based response system (IWRS). There will be unblinded team which consists of pharmacist and nurse who will give injection. All the safety assessment will be performed independently by clinical team.

Subjects will be follow-up for assessing immunity at day 28 (V3), day 60 (V4) and day 90 (V5) and for safety at day 7 (V2), day 28 (V3), day 60 (V4) and day 90 (V5).

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female age equal or more than 20 years with Thai ID cards
2. Received two doses (21-28 days apart) of Sinovac inactivated COVID-19 vaccine who will be divided according to their intervals 60-less than 90 days, 90-less than120 days and 120-180 days
3. Has provided written informed consent prior to performance of any study-specific procedure
4. No history of fever or PUI symptoms within 7 days

Exclusion Criteria:

1. Any confirmed or suspected immunosuppressive or immunodeficient state.
2. Contraindication to AZ or PF according to labelling of the products
3. History of COVID infection within 3 months period
4. Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
GMT Anti-S IgG at baseline and after vaccination | Day 0, Day 28, Day 60 and Day 90
  GMT Anti-S IgG at baseline and after vaccination at day 28, day 60 and day 90
GMFR changed from baseline in anti-S IgG GMT after vaccination | Day 28, Day 60 and Day 90
  GMFR changed from baseline in anti-S IgG GMT at 28,60 and 90 days after vaccination
Anti-S IgG Seroresponses changed from baseline after vaccination | Day 28, Day 60 and Day 90
  Frequency and percentage of participants with seroresponses in anti-S IgG titer as defined by (1) a ≥ 4-fold increase from baseline at 28, 60 and 90 days after vaccination (2) a ≥ 10-fold increase from baseline at 28,60 and 90 days after vaccination
GMT against SARS-Cov-2 pseudovirus (PVNT) Neutralizing antibody titer 50 at baseline and after vaccination | Day 0, Day 28 and Day 90
  GMT against SARS-Cov-2 pseudovirus (PVNT) Neutralizing antibody titer 50 at baseline and after vaccination at day 28 and day 90
GMFR changed from baseline in NT50 against SARS-CoV-2 pseudovirus after vaccination | Day 28 and Day 90
  GMFR changed from baseline in NT50 against SARS-CoV-2 pseudovirus at 28 and 90 days vaccination
Frequency of solicited reportable local adverse event after vaccination | Day 0 through Day 7
  Frequency and percentage of solicited reportable local adverse events (pain or tenderness, erythema, swelling or induration) of vaccination
Frequency of solicited reportable systemic adverse event after vaccination | Day 0 through Day 7
  Frequency and percentage of solicited reportable systemic adverse events (fever, headache, fatigue or malaise, myalgia, arthralgia, nausea or vomitting) of vaccination
Frequency of all unsolicited AEs | Day 0 through Day 28
  Frequency and percentage of all unsolicited AEs
Frequency of SAEs | Day 0 through Day 90
  Frequency and percentage of SAEs throughout the entire study period

SECONDARY OUTCOMES:
NT50 GMT against SARS-Cov-2 by micro neutralization assay at baseline and day 28 and day 90 after vaccination | Day 0, Day 28 and Day 90
  NT50 GMT against SARS-Cov-2 by micro neutralization assay at baseline and day 28 and 90 after vaccination
GMFR changed from baseline in NT50 against SARS-CoV-2 (micro NT Delta/WT NA) at 28 and 90 days after vaccination among those positives by PNT assay | Day 28 and Day 90
  GMFR changed from baseline in NT50 against SARS-CoV-2 (micro NT Delta/WT NA) at 28 and 90 days after vaccination among those positives by PNT assay
NT50 seroresponses against SARS-CoV-2 using micro NT changed from baseline at 28 and 90 days after vaccination among those positive by PVNT assay | Day 28 and Day 90
  Frequency and percentage of participants with NT50 seroresponses against SARS-CoV-2 using micro NT as defined by (1) a ≥ 4-fold increase from baseline at 28 and 90 days after vaccination compare to baseline among those positive by PVNT assay

OTHER OUTCOMES:
S protein-specific T cells response at baseline, 28 days after vaccination given at different intervals | Day 28
  Frequency and percentage of S protein-specific T cells response elicited by each of the regimens as measured by QuantiFERON at baseline and 28 days after vaccination
Seroresponse against SARS-CoV-2 pseudovirus towards Omicron strains at baseline, 28 and 90 days after vaccination | Day 0, 28 and 90
  Frequency and percentage of subjects with % inhibition response at 1:80 dilution against SARS-CoV-2 pseudovirus as defined by more than 50% and 68% inhibition towards Omicron strains
NT50 GMT against SARS-Cov-2 pseudovirus (pVNT) Omicrron strain at baseline 28 and 90 days after vaccination | Day 0, 28 and 90
  NT50 GMT against SARS-Cov-2 pseudovirus (pVNT) Omicrron strain at baseline 28 and 90 days after vaccination
GMFR changed from baseline in NT50 against SARS-CoV-2 pseudovirus (pVNT), Omicron strain at 28 and 90 days after vaccination | Day 28, 90
  GMFR changed from baseline in NT50 against SARS-CoV-2 pseudovirus (pVNT), Omicron strain at 28 and 90 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, MD, Study Chair — Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University; Atibordee Meesing, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University; Romanee Chaiwarith, MD,MHS, Principal Investigator — Faculty of Medicine, Chiang Mai University; Sarunyou Chusri, MD,PhD, Principal Investigator — Faculty of Medicine, Prince of Songkla University; Sira Nanthapisal, MD,PhD, Principal Investigator — Faculty of Medicine, Thammasat University; Suppachok Kirdlarp, MD, Principal Investigator — Chakri Naruebodindra Medical Institute, Faculty of Medicine Ramathibodi hospital,Mahidol University; Suvimol Niyomnaitham, MD,PhD, Principal Investigator — Mahidol University; Sarawut Siwamogsatham, MD, Principal Investigator — Chulalongkorn University
Locations (7):
- Thailand (7):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok
  - Faculty of Medicine Chulalongkorn University, Pathum Wan, Bangkok
  - Faculty of Medicine Thammasat University, Khlong Luang, Changwat Pathum Thani
  - Chakri Naruebodindra Medical Institute, Faculty of Medicine Ramathibodi hospital, Mahidol University, Bang Phli, Changwat Samut Prakan
  - Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Faculty of Medicine, Khon Kaen University, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
data or left over specimen will be shared for future study ONLY subject who consent allow using their data/specimens. Sharing will be done without personnel identification
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: as document attach when completed study in NCT clinicaltrials.gov